CLINICAL TRIAL: NCT04509934
Title: The Effect of Connective Tissue Manipulation on General Health and Emotional Status in Women With Primary Dysmenorrhea: Long-Term Follow-Up
Brief Title: The Effect of Connective Tissue Manipulation on General Health and Emotional Status in Women With Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Aybike Senel, Research Assistant, Sub-investigator, Physiotherapist, MSc, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12
Record Dates: First submitted 2020-07-14; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Primary Dysmenorrhea
Keywords: primary dysmenorrhea; pain; women; connective tissue manipulation; longterm follow up
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistical analyses will be performed by the statistics specialist that does not know anything about the methodology of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Connective Tissue Manipulation was performed to participants in Group 1, starting at the end of the menstrual cycle, 5 days a week and for 1 cycle (approximately 3 weeks) until the beginning of the next period.
  Interventions: Other: Connective Tissue Manipulation
- Group 2 (Active Comparator): In Group 2, Connective Tissue Manipulation was started with the completion of menstrual cycle performed to participants for 5 days a week and until the other menstrual cycles. At the end of the menstrual cycle, it was restarted and a total of 2 cycles were applied until the second menstrual cycle started (approximately 6 weeks).
  Interventions: Other: Connective Tissue Manipulation

INTERVENTIONS:
Other: Connective Tissue Manipulation — The position of the patients during treatment sessions was sitting with the hips and knees at 90° flexion and feet supported, arms relaxed on the thighs, back naked and straight, allowing optimal tension of the connective tissue. The CTM procedure consisted of treating 3 sections in the back. These sections were basic (sacral and lumbar regions), lower thoracic (L1 through T7) and anterior pelvic. All sessions were ended with bilateral long strokes to the iliac crest and subcostal regions. The physiotherapist applied strokes bilaterally by her middle finger of the right or left hand to the defined zones of the mentioned sections in the back. The treatment started from the basic section, and progress to other regions was decided according to the vascular reaction of the connective tissue. Each session lasted for 5 to 20 minutes, depending on the extent of the treated area.

SUMMARY:
The purpose of this study was to reveal the effects of connective tissue manipulation (CTM) on pain severity, fatigue, sleep quality, general health status, systemic symptoms, anxiety and depression in women with primary dysmenorrhoea and to determine the effect of treatment time on recovery in a longterm period. Our primary outcome was intensity of menstrual pain. Secondary outcomes were intensity of sleep disturbance, fatigue, depression and anxiety status, general health and premenstrual symptoms.

DETAILED DESCRIPTION:
The purpose of this study was to reveal the effects of CTM on pain severity, fatigue, sleep quality, general health status, systemic symptoms, anxiety and depression in women with primary dysmenorrhoea and to determine the effect of treatment time on recovery in a longterm period. Our primary outcome was intensity of menstrual pain. Secondary outcomes were intensity of sleep disturbance, fatigue, depression and anxiety status, general health and premenstrual symptoms. The participants included to this study were randomised into two groups with simple randomisation method. CTM was performed to participants in both groups included the basic region (Sacral and lumbar), lower thoracic (between T12-T7) and anterior pelvic regions. In Group 1, starting at the end of the menstrual cycle, CTM was applied for 5 days a week and for 1 cycle (approximately 3 weeks) until the beginning of the next period. Participants in the Group 2 CTM was started with the completion of menstrual cycle, 5 days a week and until the other menstrual cycles. At the end of the menstrual cycle, it was restarted and a total of 2 cycles were applied until the second menstrual cycle started (approximately 6 weeks). Both short and long strokes were used during manipulation. Each stroke was repeated for three times first on the right and then on the left side of all manipulated regions. All sessions were ended with bilateral long strokes to the iliac crest and subcostal regions. The treatment was started from the basic region and proceeded to other regions according to the vascular reaction of the connective tissue. Each session lasted 5 to 20 minutes, depending on the size of the treated region. During manipulation, the pad of the middle finger was in contact with the patient's skin. The finger was placed on the skin at 45° angle with distal interphalangeal joint in flexion and moved to cause traction. During back treatment, the participant was asked to sit erect, with hips, knees, and ankles at 90° flexion and thighs and feet are fully supported. During the treatment of anterior pelvic region, the patient was in a supine position with pillows placed under the head and knees. Treatment was performed by a trained physiotherapist. The participants' intensity of pain, fatigue and sleep quality were assessed with Visual Analogue Scale. Depressive symptoms and anxiety status, general health and premenstrual symptoms were assessed with Beck Depression Inventory, Beck Anxiety Inventory, General Health Questionnaire and Premenstrual Syndrome Scale, respectively. All measurements were repeated 5 times; baseline, after the first menstruation following the intervention period, 3th, 6th and 12th months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being in a age range 18-30
* Diagnosed with Primary Dysmenorrhea by a gynecologist
* Having a regular menstrual cycle (28±7 days)
* Being nulliparous
* Having menstrual pain intensity above 5cm according to Visual Analog Scale

Exclusion Criteria:

* Having gastrointestinal, urogynecologic, or psychiatric disease, other chronic pain syndromes
* Having a positive pregnancy test
* History of pelvic surgery
* Usage of oral contraceptives or antidepressants for at least 3 months
* Having irregular menstrual cycles (defined as lasting<21or>35 days)
* Having a history or an ultrasonographic observation of pathological conditions indicating secondary dysmenorrhea

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | baseline (first assessment) and 3th, 6th and 12th months after treatment
  Intensity of menstrual pain was evaluated by a 0- to 10-cm Visual Analog Scale (VAS), where "0" point indicated "no pain" and "10" indicated "unbearable pain."
Visual Analogue Scale | 3th month after treatment
  Intensity of menstrual pain was evaluated by a 0- to 10-cm Visual Analog Scale (VAS), where "0" point indicated "no pain" and "10" indicated "unbearable pain."
Visual Analogue Scale | 6th month after treatment
  Intensity of menstrual pain was evaluated by a 0- to 10-cm Visual Analog Scale (VAS), where "0" point indicated "no pain" and "10" indicated "unbearable pain."
Visual Analogue Scale | 12th month after treatment
  Intensity of menstrual pain was evaluated by a 0- to 10-cm Visual Analog Scale (VAS), where "0" point indicated "no pain" and "10" indicated "unbearable pain."

SECONDARY OUTCOMES:
Visual Analogue Scale | baseline (first assessment)
  Intensity of sleep disturbance was evaluated by a 0- to 10-cm Visual Analog Scale (VAS), where "0" point indicated "no sleep disturbance" and "10" indicated "unbearable disturbance."
Visual Analogue Scale | 3th month after treatment
  Intensity of sleep disturbance was evaluated by a 0- to 10-cm Visual Analog Scale (VAS), where "0" point indicated "no sleep disturbance" and "10" indicated "unbearable disturbance."
Visual Analogue Scale | 6th month after treatment
  Intensity of sleep disturbance was evaluated by a 0- to 10-cm Visual Analog Scale (VAS), where "0" point indicated "no sleep disturbance" and "10" indicated "unbearable disturbance."
Visual Analogue Scale | 12th month after treatment
  Intensity of sleep disturbance was evaluated by a 0- to 10-cm Visual Analog Scale (VAS), where "0" point indicated "no sleep disturbance" and "10" indicated "unbearable disturbance."
Visual Analogue Scale | baseline (first assessment)
  Fatigue status of the participants during dysmenorrhea was evaluated using a 10 cm VAS. Participants were asked to mark the severity of the fatigue they felt on the 10 cm line, which wrote an unbearable fatigue on one end and the other end no fatigue.
Visual Analogue Scale | 3th month after treatment
  Fatigue status of the participants during dysmenorrhea was evaluated using a 10 cm VAS. Participants were asked to mark the severity of the fatigue they felt on the 10 cm line, which wrote an unbearable fatigue on one end and the other end no fatigue.
Visual Analogue Scale | 6th month after treatment
  Fatigue status of the participants during dysmenorrhea was evaluated using a 10 cm VAS. Participants were asked to mark the severity of the fatigue they felt on the 10 cm line, which wrote an unbearable fatigue on one end and the other end no fatigue.
Visual Analogue Scale | 12th month after treatment
  Fatigue status of the participants during dysmenorrhea was evaluated using a 10 cm VAS. Participants were asked to mark the severity of the fatigue they felt on the 10 cm line, which wrote an unbearable fatigue on one end and the other end no fatigue.
Beck Depression Inventory | baseline (first assessment)
  Beck Depression Inventory which is self-administrated questionnaire was used to determine depressive symptoms during the menstrual periods of the participants. The inventory includes 21 questions and is scored by adding the scores of each question, which are scored between 0 and 3. Lower scores indicate less depressive symptoms, while higher scores show more depressive symptoms
Beck Depression Inventory | 3th month after treatment
  Beck Depression Inventory which is self-administrated questionnaire was used to determine depressive symptoms during the menstrual periods of the participants. The inventory includes 21 questions and is scored by adding the scores of each question, which are scored between 0 and 3. Lower scores indicate less depressive symptoms, while higher scores show more depressive symptoms
Beck Depression Inventory | 6th month after treatment
  Beck Depression Inventory which is self-administrated questionnaire was used to determine depressive symptoms during the menstrual periods of the participants. The inventory includes 21 questions and is scored by adding the scores of each question, which are scored between 0 and 3. Lower scores indicate less depressive symptoms, while higher scores show more depressive symptoms
Beck Depression Inventory | 12th month after treatment
  Beck Depression Inventory which is self-administrated questionnaire was used to determine depressive symptoms during the menstrual periods of the participants. The inventory includes 21 questions and is scored by adding the scores of each question, which are scored between 0 and 3. Lower scores indicate less depressive symptoms, while higher scores show more depressive symptoms
Beck Anxiety Inventory | baseline (first assessment)
  Anxiety experienced by participants during menstrual periods was measured using Beck Anxiety Inventory (BAI). Each item is rated on a 4-point scale reflecting the degree to which each symptom disturbs participants; the answer options range from 0 (not at all) to 3 (severely, I could barely stand it). With higher scores indicating more severe anxiety.
Beck Anxiety Inventory | 3th month after treatment
  Anxiety experienced by participants during menstrual periods was measured using Beck Anxiety Inventory (BAI). Each item is rated on a 4-point scale reflecting the degree to which each symptom disturbs participants; the answer options range from 0 (not at all) to 3 (severely, I could barely stand it). With higher scores indicating more severe anxiety.
Beck Anxiety Inventory | 6th month after treatment
  Anxiety experienced by participants during menstrual periods was measured using Beck Anxiety Inventory (BAI). Each item is rated on a 4-point scale reflecting the degree to which each symptom disturbs participants; the answer options range from 0 (not at all) to 3 (severely, I could barely stand it). With higher scores indicating more severe anxiety.
Beck Anxiety Inventory | 12th month after treatment
  Anxiety experienced by participants during menstrual periods was measured using Beck Anxiety Inventory (BAI). Each item is rated on a 4-point scale reflecting the degree to which each symptom disturbs participants; the answer options range from 0 (not at all) to 3 (severely, I could barely stand it). With higher scores indicating more severe anxiety.
General Health Questionnaire | baseline (first assessment)
  General Health Questionnaire was used to determine the health status of the participants during their menstrual periods. A 28 item scaled version-assesses somatic symptoms, anxiety, and insomnia, social dysfunction and severe depression. Likert's numbering method (as 0, 1, 2, and 3) was utilized. It means that scores higher than 6 in subscales and totally higher than 22 indicates chronic symptoms.
General Health Questionnaire | 3th month after treatment
  General Health Questionnaire was used to determine the health status of the participants during their menstrual periods. A 28 item scaled version-assesses somatic symptoms, anxiety, and insomnia, social dysfunction and severe depression. Likert's numbering method (as 0, 1, 2, and 3) was utilized. It means that scores higher than 6 in subscales and totally higher than 22 indicates chronic symptoms.
General Health Questionnaire | 6th month after treatment
  General Health Questionnaire was used to determine the health status of the participants during their menstrual periods. A 28 item scaled version-assesses somatic symptoms, anxiety, and insomnia, social dysfunction and severe depression. Likert's numbering method (as 0, 1, 2, and 3) was utilized. It means that scores higher than 6 in subscales and totally higher than 22 indicates chronic symptoms.
General Health Questionnaire | 12th month after treatment
  General Health Questionnaire was used to determine the health status of the participants during their menstrual periods. A 28 item scaled version-assesses somatic symptoms, anxiety, and insomnia, social dysfunction and severe depression. Likert's numbering method (as 0, 1, 2, and 3) was utilized. It means that scores higher than 6 in subscales and totally higher than 22 indicates chronic symptoms.
Premenstrual Syndrome Scale | baseline (first assessment)
  Premenstrual Syndrome Scale was used to measure the severity of the participants' premenstrual symptoms. The lowest possible total score is 44 points and the highest is 220. High PMSS score indicates more severe premenstrual symptoms.
Premenstrual Syndrome Scale | 3th month after treatment
  Premenstrual Syndrome Scale was used to measure the severity of the participants' premenstrual symptoms. The lowest possible total score is 44 points and the highest is 220. High PMSS score indicates more severe premenstrual symptoms.
Premenstrual Syndrome Scale | 6th month after treatment
  Premenstrual Syndrome Scale was used to measure the severity of the participants' premenstrual symptoms. The lowest possible total score is 44 points and the highest is 220. High PMSS score indicates more severe premenstrual symptoms.
Premenstrual Syndrome Scale | 12th month after treatment
  Premenstrual Syndrome Scale was used to measure the severity of the participants' premenstrual symptoms. The lowest possible total score is 44 points and the highest is 220. High PMSS score indicates more severe premenstrual symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Nesrin Yağcı, PT, Prof, Study Chair — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yagci N, Senel A, Atalay OT, Akman TC, Can OK. Long-Term Follow-Up Result of Connective Tissue Manipulation in Young Women with Primary Dysmenorrhea: Different Intervention Durations. Reprod Sci. 2023 Jul;30(7):2198-2209. doi: 10.1007/s43032-023-01172-5. Epub 2023 Jan 30. PMID 36717461